CLINICAL TRIAL: NCT06804863
Title: Monitoring and Timely Intervention of Regret Emotion After Thyroidectomy in Low-Risk Papillary Thyroid Cancer Patients: A Multicenter, Randomized, Controlled Trial
Brief Title: Regret Emotion After Thyroidectomy in Low-Risk Papillary Thyroid Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xinyi Wang, Dr, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WestChinaH20220423
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer; Regret
Keywords: Papillary thyroid cancer; regret; active intervention; prognosis
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: The REDCap randomization module will be used, and block randomization will be computer-generated with block sizes of 6 and 9, in a 1:1 ratio, to allocate patients to either the intervention or control group. The allocation sequence will be concealed, and the randomized results will be extracted by an independent data collection team. If intervention group patients need to complete the QoL scale, after completion, the doctor from the department corresponding to the factor with the highest score (i.e., the factor most closely related to the patient's regret state) will receive an SMS notification and will be required to contact the patient by phone or SMS within 24 hours to provide the intervention. If contact is not established within 24 hours of the intervention phase, the research participant will call the patient up to two times to clarify the reason.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervening in patients with postoperative regret emotion. (Experimental): For the worst postoperative quality of life factors reported by patients, specialized doctors will provide immediate guidance and management via SMS or phone.
  Interventions: Behavioral: Postoperative Regret Reduction through Immediate Quality of Life Intervention
- Only the patients' postoperative regret levels and quality of life scores will be collected. (No Intervention): Only the patients' postoperative regret levels and quality of life scores will be collected, without any additional interventions.

INTERVENTIONS:
Behavioral: Postoperative Regret Reduction through Immediate Quality of Life Intervention — Immediate intervention of the major impaired quality of life factors postoperatively to reduce patients' postoperative regret.
  Arms: Intervening in patients with postoperative regret emotion.

SUMMARY:
This randomized, active-controlled, non-inferiority trial is scheduled to begin in May 2025 and will continue until June 2027. Inclusion criteria: (1) Patients with low-risk papillary thyroid cancer without lymph node metastasis who have undergone thyroid surgery (including both laparoscopic and open surgery) at the Department of Thyroid Surgery, West China Hospital, Sichuan University, (2) Aged between 18 and 90 years, (3) Chinese-speaking, (4) Capable of completing questionnaires and using a mobile phone and internet for intervention purposes, (5) No history of psychiatric disorders or use of psychotropic medications, (6) Voluntary participation and signing of an informed consent form. Exclusion criteria: (1) Patients with cervical lymph node metastasis, (2) Incomplete baseline data, (3) Uncontrolled chronic diseases, (4) Patients with other cancers. Online outpatient follow-up will be conducted by doctors from the Department of Thyroid Surgery at West China Hospital. One study participant will contact the patient, introduce the study, and obtain the informed consent form from willing participants. The research team members responsible for patient contact, registration, and randomization include the principal investigator, study coordinator, and specially trained research assistants. The management of the intervention group patients will be carried out by doctors from the corresponding departments. According to the protocol, patients assigned to online visits will switch to offline visits and exit the clinical trial under the following circumstances: (1) unresolved technical issues, (2) inability to perform a comprehensive assessment, (3) patient request for withdrawal. Other cross-cutting reasons include patient requests and scheduling conflicts. Baseline data (including age, gender, ethnicity, address, occupation), tumor-related information (including tumor histology, maximum tumor diameter, capsular invasion status, number of lymph node metastases), and surgical method will be collected from the hospital's information department. Participants will be given the DRS scale upon discharge and every two months thereafter to assess their regret status. For patients with high regret (DRS score >25), a QoL scale will be further distributed to collect information about their quality of life. The REDCap randomization module will be used, and block randomization will be computer-generated with block sizes of 6 and 9, in a 1:1 ratio, to allocate patients to either the intervention or control group. The allocation sequence will be concealed, and the randomized results will be extracted by an independent data collection team. If intervention group patients need to complete the QoL scale, after completion, the doctor from the department corresponding to the factor with the highest score (i.e., the factor most closely related to the patient's regret state) will receive an SMS notification and will be required to contact the patient by phone or SMS within 24 hours to provide the intervention. If contact is not established within 24 hours of the intervention phase, the research participant will call the patient up to two times to clarify the reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with low-risk papillary thyroid cancer without lymph node metastasis who have undergone thyroid surgery,
2. Aged between 18 and 90 years,
3. Chinese-speaking,
4. Capable of completing questionnaires and using a mobile phone and internet for intervention purposes,
5. No history of psychiatric disorders or use of psychotropic medications,
6. Voluntary participation and signing of an informed consent form.

Exclusion Criteria:

1. Patients with cervical lymph node metastasis,
2. Incomplete baseline data,
3. Uncontrolled chronic diseases,
4. Patients with other cancers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Clarifying the impact of immediate intervention on patients' postoperative regret psychology. | From enrollment to the end of follow-up at 12 months
  Over a 12-month period after the start of the study, observe the declining trend of regret scores in patients who received immediate intervention compared to the control group.

SECONDARY OUTCOMES:
Main Factors Affecting Postoperative Regret in Low-Risk PTC Patients | From enrollment to the end of follow-up at 12 months
  Over a 12-month period after the start of the study, evaluate patients' quality of life in different aspects following thyroid cancer surgery at each time point using the thyroid cancer-specific Quality of Life (QoL) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China